CLINICAL TRIAL: NCT06021938
Title: Alleviating Persistent Dyspnea in Amyotrophic Lateral Sclerosis Patients Treated With Non-Invasive Ventilation Through Immersive Virtual Reality
Acronym: RVI-SLA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP230974
Record Dates: First submitted 2023-08-25; First posted 2023-09-01 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Persistent Dyspnea; Non-Invasive Ventilation; Immersive Virtual Reality
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients starting with RVI (Active Comparator): Patients will begin by wear a virtual reality headset (GAMIDA®) and headphones (Bose®). A tablet (Samsung®) equipped with "Healthy Mind" software will allow patients to live a 360° visual and auditory 3D experience via Bluetooth connection. After that patients will be handed a smartphone with the Spotify® application to listen to music. Patients will wear headphones.
  Interventions: Device: Immersive virtual reality (IVR) & Music therapy
- Patients starting with music therapy (Active Comparator): Patients will begin by handed a smartphone with the Spotify® application to listen to music. Patients will wear headphones. After that patients will wear a virtual reality headset (GAMIDA®) and headphones (Bose®). A tablet (Samsung®) equipped with "Healthy Mind" software will allow patients to live a 360° visual and auditory 3D experience via Bluetooth connection.
  Interventions: Device: Immersive virtual reality (IVR) & Music therapy

INTERVENTIONS:
Device: Immersive virtual reality (IVR) & Music therapy — The patient will be offered a digital therapy session based on immersive virtual reality (IVR) and a music therapy session, 60 minutes apart. The IVR session will be based on medical hypnosis (GAMIDA®) and the music therapy session will be based on the choice of music the patient wishes. Each session will last 15 minutes. Patients will start either with the medical hypnosis session by IVR or with the music session depending on the randomization carried out before the start of the study. The random order will be provided by software (CleanWeb).

SUMMARY:
The evolution of amyotrophic lateral sclerosis (ALS) is marked by dyspnea, anxiety and pain, major determinants of suffering induced by this disease. The only palliative treatment for respiratory failure is non-invasive ventilation (NIV), which compensates failing respiratory muscles and relieves dyspnea, improves quality of life and increases life expectancy. In ALS patients, the persistence of dyspnea outside of NIV sessions has highlighted the need for therapeutic alternatives in the treatment of persistent dyspnea, including immersive virtual reality (IVR) and auditory distraction through music (music therapy). This study evaluates the effect of IVR on respiratory discomfort in ALS patients with persistent dyspnea treated with NIV.

DETAILED DESCRIPTION:
The evolution of amyotrophic lateral sclerosis (ALS) is marked by dyspnea, anxiety and pain, major determinants of suffering induced by this disease. The only palliative treatment for respiratory failure is non-invasive ventilation (NIV), which compensates failing respiratory muscles and relieves dyspnea, improves quality of life and increases life expectancy. In ALS patients, the persistence of dyspnea outside of NIV sessions has highlighted the need for therapeutic alternatives in the treatment of persistent dyspnea, including immersive virtual reality (IVR) and auditory distraction through music (music therapy). The objective of this study is to evaluate the effect of IVR on respiratory discomfort (scale A1 of the Multidimensional Dyspnea Profile (MDP) questionnaire) of patients with ALS at the stage of respiratory failure treated with NIV. This will be an open-label, monocentric, randomized, controlled cross-over clinical study. ALS patients will be recruited during their respiratory evaluation carried out as part of their usual care provided in an ambulatory setting (day care hospital) in the Pneumology Department of Pitié Salpêtrière Hospital. Eligibility criteria will be verified during this visit. If the patient meets eligibility criteria, the investigator will present the study to him using the information letter. After a period of reflection that the patient deems necessary to make his decision and after having obtained an answer to all his questions, his written consent will be collected by the investigator. The patient will then be offered a digital therapy session based on immersive virtual reality (IVR) and a music therapy session, 60 minutes apart. The IVR session will be based on medical hypnosis (GAMIDA®) and the music therapy session will be based on the choice of music that the patient wishes. Each session will last 15 minutes. Patients will start either with the medical hypnosis session by IVR or with the music session depending on the randomization carried out before the start of the study. The random order will be provided by software (CleanWeb).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Diagnosis of ALS confirmed according to the revised criteria of El Escorial
* Respiratory failure due to diaphragmatic dysfunction treated by non-invasive ventilation for more than a month
* Care provided in an ambulatory setting (day care hospital)
* Persistent dyspnea at rest ≥ 3 across a numerical scale (0 to 10) in a semi-sitting position
* Stable clinical condition, i.e., no episode of acute cardiac, respiratory and/or neurological failure leading to hospitalization in the previous 4 weeks
* Free, prior and informed written consent about the study has been obtained
* Benefiting a social security (French health insurance system)

Exclusion Criteria:

* Neurological disorders according to a neurological evaluation dating from less than one year, in particular diagnosed dementia (frontotemporal dementia, Alzheimer's disease, etc.), brain pathology (tumor, stroke, Parkinson's disease, etc.)
* Diagnosed psychiatric illness (severe depression, psychosis) or receiving antipsychotic treatment
* Acrophobia
* Claustrophobia
* Photophobia
* Hearing loss
* Visual impairment
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2026-04-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of IVR on respiratory discomfort (A1) | 15 minutes
  Evaluate the effect of IVR on respiratory discomfort (scale A1 of the MDP questionnaire) of patients with ALS at the stage of respiratory failure treated with NIV

SECONDARY OUTCOMES:
Evaluate the effect of IVR on respiratory discomfort (QS and A2) | 15 minutes
  Evaluate the effect of IVR on the sensory (scale QS of the MDP questionnaire) and emotional (scale A2 of the MDP questionnaire) components of dyspnea of patients with ALS at the stage of respiratory failure treated with NIV.
Evaluate the effect of music therapy on respiratory discomfort (QS, A1 and A2) | 15 minutes
  Evaluate the effect of music therapy on the sensory (scale QS of the MDP questionnaire), affective (scale A1 of the MDP questionnaire) and emotional (scale A2 of the MDP questionnaire) components of dyspnea of patients with ALS at the stage of respiratory failure treated with NIV.
Compare the evolutionary profile on respiratory discomfort (QS, A1 and A2) under the effect of IVR and music therapy | 15 minutes
  Compare the evolutionary profile of the sensory ( scale QS of the MDP questionnaire ) and affective ( scale A1 and A2 of the MDP questionnaire) components of dyspnea under the effect of IVR and music therapy.
Compare the effect of IVR and music therapy on the respiratory discomfort in terms of preference. | 15 minutes
  Compare the effect of IVR and music therapy on the respiratory discomfort of ALS patients treated with NIV in terms of preference through a post-exposure questionnaire after the two interventions
Evaluate the acceptability of IVR | 15 minutes
  Evaluate the effect of IVR on dyspnea in terms of acceptability by a subjective questionnaire of six questions using a 7-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie, Paris, France, France

IPD SHARING:
Plan to Share IPD: No